CLINICAL TRIAL: NCT01343810
Title: The Effect of Mindfulness-Based Stress Reduction on Sleep Quality, Stress Physiology & CVD Risk
Brief Title: Stress Reduction Training to Improve Sleep Quality, Stress Physiology & Cardiovascular Disease (CVD) Risk Markers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jeffrey M. Greeson, PhD, Duke University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00025227; 4R00AT004945-03 (NIH)
Record Dates: First submitted 2011-04-25; First posted 2011-04-28 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Stress, Psychological; Sleep; Inflammation; Cardiovascular Diseases
Keywords: Mindfulness-Based Stress Reduction; Meditation; Psychological stress; Sleep quality; Cardiovascular disease; Inflammation
MeSH Terms: conditions — Stress, Psychological; Inflammation; Cardiovascular Diseases; Sleep Initiation and Maintenance Disorders | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Meditation (Experimental): Both arms will undergo 8-weeks of Mindfulness-Based Stress Reduction (MBSR) training. The experimental arm will be randomly assigned to practice meditation immediately following the emotional stress task in the lab during the post-MBSR lab visit.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR); Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- No meditation (Active Comparator): Both arms will undergo 8-weeks of Mindfulness-Based Stress Reduction (MBSR) training. The active comparator arm will be randomly assigned to not practice meditation, but rather listen to a non-meditative audio track of equal length, immediately following the emotional stress task in the lab during the post-MBSR lab visit.
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR); Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction (MBSR) — The MBSR program consists of 8 weekly classes that last for 2.5 hours each and a commitment to daily meditation practice for the duration of the course. Classes include didactic instruction on mindfulness and its relationship to stress and health, guided meditation practices, and group discussion. Mindfulness meditation practices include awareness of breathing, awareness of emotions, body scan, mindful hatha yoga, mindful walking, mindful eating, mindful listening, and lovingkindness (metta). Participants are expected to practice formal meditation outside of class for 20-45 min per day, 6 days per week. In addition, participants are encouraged apply mindfulness to everyday activities like eating, communicating with others, and hobbies. Written materials and audio CDs with guided meditations and yoga are provided. The course also includes one full day (7-hours) of meditation on a Saturday following the 6th week of class.
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — The MBSR program consists of 8 weekly classes that last for 2.5 hours each and a commitment to daily meditation practice for the duration of the course. Classes include didactic instruction on mindfulness and its relationship to stress and health, guided meditation practices, and group discussion. Mindfulness meditation practices include awareness of breathing, awareness of emotions, body scan, mindful hatha yoga, mindful walking, mindful eating, mindful listening, and lovingkindness (metta). Participants are expected to practice formal meditation outside of class for 20-45 min per day, 6 days per week. In addition, participants are encouraged apply mindfulness to everyday activities like eating, communicating with others, and hobbies. Written materials and audio CDs with guided meditations and yoga are provided. The course also includes one full day (7-hours) of meditation on a Saturday following the 6th week of class.

SUMMARY:
The goal of this study is to better understand the potential value of reducing stress to ameliorate a cluster of biological and behavioral factors implicated in cardiovascular disease (CVD) risk. These factors include psychological distress, poor sleep quality, and exaggerated physiological responses to emotional stress. Results will be used to develop an innovative brief intervention to reduce risk for CVD by improving sleep quality, ameliorating psychological distress, and attenuating stress physiology.

DETAILED DESCRIPTION:
This study will be conducted among 200 men and women participating in 8-week Mindfulness-Based Stress Reduction (MBSR) classes at Duke Integrative Medicine in Durham, North Carolina. The central hypothesis of this NIH-funded clinical trial (R00 AT004945, PI: Greeson) is that mindfulness meditation training is associated with increased levels of mindfulness and improved cognitive-emotional functioning that, together, are associated with reduced psychological distress, improved sleep quality, and less exaggerated physiological responses to emotional stress, including blood pressure and inflammation. This study is designed to examine psychological and biological mechanisms that may explain individual differences in MBSR outcomes. This knowledge is important because it will help us better understand who is most likely to benefit from mindfulness meditation training, and why. The results from this study are expected to elucidate mechanisms underlying the mental and physical health benefits of stress reduction, which can help guide clinicians in referring the most suitable patients to local MBSR programs.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in an 8 week stress reduction training program
2. Between 18 and 65 years old
3. Generally in good health and not taking medication
4. Able to speak and read English
5. Willing to provide informed consent
6. Able to access the internet
7. Able to attend 4 study visits at Duke University Medical Center

Exclusion Criteria:

1. Younger than 18 years old/Older than 65
2. Asthma
3. Allergies
4. Arthritis
5. Autoimmune disease (Lupus)
6. Cancer
7. Cardiovascular disease, heart attack, or atherosclerosis
8. Diabetes or High Blood Sugar (>124 mg/dl)
9. Hypertension or high blood pressure (140/90 mmHg)
10. High cholesterol (>240 mg/dl)
11. Obesity (Body Mass Index >30)
12. Irritable Bowel Syndrome (IBS)
13. Mitral Valve Prolapse, or Heart Murmurs
14. Irregular Menstrual Cycles (Peri-Menopause Excluded. Menopause may be included.)
15. Skin conditions, such as eczema or psoriasis (acne may be included)
16. Sleep Apnea
17. Depression, anxiety, substance use, or any other mental health diagnosis
18. Sleep aids like Tylenol PM or Ambien on a regular basis
19. Medication for allergies or asthma on a regular basis
20. Aspirin or baby Aspirin on a regular basis
21. Oral contraceptives or birth control (women only)
22. Hormone Replacement Therapy
23. Flu shot within past 3 weeks
24. Underweight (BMI < 18.5)
25. Current smoker
26. >1 alcoholic drink/day (women)/ >2 alcoholic drinks/day (men)
27. Hospitalized within the last 3 months
28. Treated for any infections within the last 3 months
29. Current meditation practice >1x/month
30. Previously taken a Mindfulness-Based Stress Reduction (MBSR) course
31. Participation in any other research studies in the past year that involved drugs or taking blood
32. Recently donated blood. (500 cc's in last 8 wks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Sleep quality | Baseline, post-intervention (2 months), follow-up (8 months)
  Sleep quality will be assessed using 3 different methods: daily sleep diaries, questionnaires and actigraphy.
Stress physiology | Baseline, post-intervention (2 months), follow-up (8 months)
  Physiological responses to mild emotional stress (5-minute Anger Recall Task) will be assessed in the laboratory before and after participating in an 8-week Mindfulness-Based Stress Reduction (MBSR) program. During the stress testing sessions, we will take measures of heart rate, blood pressure, stress hormones, metabolism, inflammation, emotions, and mindful qualities.

SECONDARY OUTCOMES:
Mindfulness | Baseline, post-intervention (2 months), follow-up (8 months)
  Mindful qualities, including observing, describing, non-judging, non-reactivity, acting with awareness, mindfulness, self-kindness, and common humanity.
Health-related quality of life | Baseline, post-intervention (2 months), follow-up (8 months)
  Global health rating; physical functioning; fatigue; satisfaction with social role; pain intensity and pain-related interference with daily activities.
Negative Affect | Baseline, post-intervention (2 months), follow-up (8 months)
  Anxiety; anger; depressive symptoms.
Cognitive functioning | Baseline, post-intervention (2 months), follow-up (8 months)
  Cognitive abilities and concerns, including attention, concentration, memory, organization, and clarity of thinking.
Emotion regulation | Baseline, post-intervention (2 months), follow-up (8 months)
  Rumination; avoidance; suppression; reappraisal.
Stress-related physical symptoms | Baseline, post-intervention (2 months), follow-up (8 months)
  Common physical symptoms associated with stress, including muscle tension, gastrointestinal complaints, headaches, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Greeson, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Integrative Medicine, Durham, North Carolina, United States